CLINICAL TRIAL: NCT04036526
Title: Randomized Double-blind Placebo-controlled Comparative Research of Potency and Safety of a GamLPV, a Live Intranasal Bordetella Pertussis Vaccine, Using Two Dosing Schedules and Methods of Application in Healthy Human Volunteers
Brief Title: A Phase 1/2 Clinical Trial of a GamLPV, a Live Intranasal Bordetella Pertussis Vaccine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GamLPV-02
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Whooping Cough
Keywords: Bordetella pertussis; Live vaccine; Immunological factors; antibody response; cell immune response; whooping cough
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Intervention Model Description: Present clinical trial is a randomized placebo-controlled study for selection of dosing schedules and application methods of GamLPV, a live intranasal Bordetella pertussis vaccine. The study is blinded for volunteers.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Drop method (Experimental): Group 1 will receive vaccine/placebo by drop method.
  Interventions: Biological: Vaccine GamLPV; Other: Placebo
- Group 2 Nasal actuator (Experimental): Group 2 will receive vaccine/placebo with nasal actuator.
  Interventions: Biological: Vaccine GamLPV; Other: Placebo

INTERVENTIONS:
Biological: Vaccine GamLPV — live intranasal vaccine for whooping cough prevention
  Other Names: live intranasal Bordetella pertussis vaccine
Other: Placebo — Placebo

SUMMARY:
The study should be leaded as a randomized double-blind placebo-controlled comparative research of potency and safety of a GamLPV, a live intranasal Bordetella pertussis vaccine, using two dosing schedules and methods of application in healthy human volunteers.

The study contains three periods: screening, inpatient hospitalization and follow-up.

DETAILED DESCRIPTION:
Subjects are divided into two groups - 25 volunteers in each group. Group 1 will receive vaccine/placebo by drop method. Group 2 will receive vaccine/placebo with nasal actuator. After 60 days both groups will repeatedly receive the same dose of vaccine/placebo by the same methods of application. In each group there are 5 volunteers given placebo.

Monitoring examination of volunteers is carrying out during 60 days after first and second vaccination.

Each group (25 persons) shall be divided into three cohorts (5, 7 and 13 persons). The arm that will receive the drug/ placebo by the dripping method comprises cohorts 1, 3, and 5, and the arm that will receive the drug using the applicator comprises cohorts 2, 4, and 6. Initially, the first and second cohorts (of 5 volunteers each) will be included into the study, respectively.

The main purpose of this study is selection of methods of applications and dosing schedules of GamLPV, a live intranasal Bordetella pertussis vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 40 (inclusively);
2. Healthy verified diagnosis according to standard clinical, laboratory and instrumental examination methods (no somatic disorder of the gastro-intestinal tract (GIT), liver, kidneys, cardiovascular system (CVS), infectious, hematological diseases, cancers (including if the preliminary standard clinical laboratory tests did not reveal any diseases);
3. BMI froim 18 to 30 kg/m2 (inclusively);
4. Consent to use of reliable birth control methods during the test period and for 3 months thereafter (a condom with spermicide);
5. Signed FactSheet and Informed Consent to Participation in the Study.
6. No specific IgM to the pertussis agent (negative IFA finding according to manufacturer's instruction for the anti-pertussis antibody detection test system);
7. Specific anti-pertussis IgG ≤ 45 EU/ml
8. No B.pertussis DNA in nasopharyngeal swabs (based on RT-PCR).

Exclusion Criteria:

1. Whooping cough in past medical history
2. Vaccination against whooping cough over the past decade
3. Any other anti-infective immunization during last year
4. Any medical condition (renal diseases, hepatic disorders, haematological malignancies, malignant neoplasms and other diseases) which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
5. Vaccine-associated diseases or clinically significant vaccinal reactions in medical history
6. Clinically significant abnormal laboratory values at the discretion of the investigator
7. Positive results of HIV, hepatitis B or C
8. Use of narcotic drugs and/or a history of drug/alcohol abuse
9. Allergic diseases in medical history (in particular drug reaction and food allergy)
10. The subject has donated blood/plasma or suffered from blood loss of at least 450 ml (1 unit of blood) within 6 weeks prior to screening
11. Current participation in any other clinical trial
12. Inability to adhere to the protocol
13. Acute infectious diseases within 4 weeks prior to screening
14. Wheezing on the results of peakflowmetry
15. Significant ECG changes
16. Pregnancy or lactation (for female volunteers)
17. Systolic blood pressure less than 90 mmHg or over than 130 mmHg; diastolic blood pressure less than 60 mmHg or over 90 mmHg
18. Heart rate less than 60 bpm or more than 90 bpm
19. Specific anti-pertussis IgG ≥ 45 EU/ml
20. The presence of B.pertussis DNA in nasopharyngeal swabs (based on RT-PCR).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-05-29 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
methods of applications | the total Time Frame is 140 days after the vaccination
  selection of methods of applications of GamLPV, a live intranasal Bordetella pertussis vaccine (drop method or nasal actuator is important for vaccination)
dosing schedules | the total Time Frame is 140 days after the vaccination
  selection of dosing schedules of GamLPV, a live intranasal Bordetella pertussis vaccine (repeated administration in 60 days)

SECONDARY OUTCOMES:
specific antibody response to B.pertussis | the total Time Frame is 140 days after the vaccination
  Evaluation of the antibody response after single and double intranasal vaccine administration in healthy volunteers with nasal actuator and by drop method compared to placebo. Detection of antibody level (IgG and IgA) in blood serum and nasopharyngeal aspirates in healthy human volunteers by ELISA.
cell immune responses to B.pertussis | the total Time Frame is 140 days after the vaccination
  Evaluation of cell immune response parameters after single and double intranasal vaccine administration in healthy volunteers with nasal actuator and by drop method compared to placebo. Detection of induced INF- γ and IL-17 quantity in PBMC supernatant (by ELISA).
dynamics of bacteria generation in nasopharynx of human volunteers | the total Time Frame is 140 days after the vaccination
  Evaluation of bacterial load in oropharynx/nasopharynx over time after single and double intranasal vaccine administration in healthy volunteers with nasal actuator and by drop method (B.pertussis DNA detection by RT-PCR method in nasopharyngeal swabs)
Comparative assessment of immunogenicity | the total Time Frame is 140 days after the vaccination
  Comparative analysis of GamLPV immunogenicity after single and double intranasal vaccine administration in healthy volunteers with nasal actuator and by drop method (by antibody response evaluation by ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Rusanova, Principal Investigator — Infectious Disease Clinical Hospital No. 1 of the Moscow Healthcare Department
Locations (1):
- Infectious Disease Clinical Hospital No. 1 of the Moscow Healthcare Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided